CLINICAL TRIAL: NCT07381452
Title: Effects of Virtual Reality-Enhanced Rehabilitation on Cognitive Recovery in Acute Post-Stroke Patients: a Pilot Study
Brief Title: Virtual Reality-Enhanced Rehabilitation for Cognitive Recovery in Acute Post-Stroke Patients: Pilot Study
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tadeja Hernja Rumpf (Other)
Responsible Party: Sponsor-Investigator, Tadeja Hernja Rumpf, Principal Investigator, University Medical Centre Maribor
Organization: University Medical Centre Maribor (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UKC-MB-KME-3/24; IRP-2021/02-08 (Other Grant/Funding Number: UKC Maribor)
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Stroke Intervention; Rehabilitation Exercise; Cognitive Assessment
Keywords: virtual reality; stroke rehabilitation; cognition; acute phase

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to the experimental group (VR training in addition to CRT) or the control group (only CRT) using sealed envelopes with group tasks in numerical sequence.
Who Masked: Investigator
Masking Description: Therapists who will evaluate participants with scales will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR + CRT (Virtual reality-enhanced rehabilitation plus Conventional rehabilitation therapy) (Experimental): The experimental group will receive physiotherapy and occupational therapy (manual therapy techniques, passive and active-assisted mobilisation, scapular mobilisation, and task-specific training such as horizontally moving an object across a surface), ten sessions over two weeks of 60 minutes per session and an additional 15 minutes of virtual-reality (VR) training per session using the Bimeo PRO system (Kinestica d.o.o., Slovenia) in a unimanual, two-dimensional configuration on a flat surface, with continuous therapist supervision.
  Interventions: Behavioral: Virtual reality-enhanced rehabilitation; Other: Conventional rehabilitation therapy (CRT)
- CRT (Conventional rehabilitation therapy) (Active Comparator): The control group will receive 10 sessions over 2 weeks of physiotherapy and occupational therapy (manual therapy techniques, passive and active-assisted mobilisation, scapular mobilisation, and task-specific training, such as moving an object horizontally across a surface), each lasting 60 minutes.
  Interventions: Other: Conventional rehabilitation therapy (CRT)

INTERVENTIONS:
Behavioral: Virtual reality-enhanced rehabilitation — Dose of practice and difficulty: In each VR session, participants will perform two tasks, completing one trial of each-a memory task and a meal-preparation task -with no within-session repetitions. Over ten sessions, participants will complete 10 trials of each task (30 in total). Task difficulty will be fixed and identical for all participants throughout the intervention (no automatic progression or therapist-driven difficulty changes). Adherence, tolerability, and adverse events: Participants will be scheduled to complete the prescribed VR dose (10 sessions; 150 minutes total). Adherence will be recorded at each session. Serious adverse events are not expected; all adverse events will be actively monitored and documented.
  Arms: VR + CRT (Virtual reality-enhanced rehabilitation plus Conventional rehabilitation therapy)
Other: Conventional rehabilitation therapy (CRT) — Physiotherapy and occupational therapy: manual therapy techniques, passive and active-assisted mobilisation, scapular mobilisation, and task-specific training, such as horizontally moving an object across a surface, 60 minutes per session.

SUMMARY:
Post-stroke rehabilitation is essential for maximising motor recovery. Virtual reality (VR) is emerging as a promising adjunct to conventional therapy (CRT), potentially enhancing upper limb motor outcomes. The goal of the study is to investigate the impact of virtual reality rehabilitation compared to conventional rehabilitation therapy on cognitive function and activities of daily living in patients with acute stroke.

DETAILED DESCRIPTION:
The investigators will conduct a prospective randomised single- blind pilot controlled trial to evaluate the efficacy of VR-based rehabilitation with the Bimeo PRO system on cognitive function and activities of daily living in patients with acute stroke. Participants will be randomly assigned to a two-week VR training program combined with conventional therapy (experimental group) or to conventional therapy alone (control group).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* First-ever acute stroke, occurring <7 days before therapy start
* Cognitive impairment on admission (Mini-Mental State Examination score < 24
* Ability to understand and perform virtual reality (VR) tasks.

Exclusion Criteria:

* Severe cognitive impairment that precludes following instructions.
* Aphasia or severe visual/hearing impairment that prevents meaningful participation.
* End-stage/terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
The Mini-Mental State Examination (MMSE) | Change from baseline to 2 weeks (end of intervention)
  It is a widely used screening tool for global cognitive function. It evaluates orientation, immediate registration and short-term recall, attention and calculation, and language and praxis. The total score ranges from 0 to 30, and scores below 24 are commonly interpreted as suggestive of cognitive impairment.
The Barthel Index (BI) | Change from baseline to 2 weeks (end of intervention)
  The Barthel Index (BI) evaluates an individual's level of independence and mobility in activities of daily living (ADLs), including feeding, bathing, grooming, dressing, bowel and bladder control, toileting, transfers, walking/ambulation, and stair climbing. It also helps determine the degree of assistance required for care.

SECONDARY OUTCOMES:
The National Institutes of Health Stroke Scale (NIHSS) | Change from baseline to 2 weeks (end of intervention)
  The NIHSS is a comprehensive assessment tool used to evaluate stroke severity. The scale generates scores ranging from 0 (denoting the absence of deficits) to 46 (signifying severe impairment).
The Modified Rankin Scale (mRS) | Change from baseline to 2 weeks (end of intervention)
  The Modified Rankin Scale (mRS) is a widely utilised and reliable functional assessment tool in clinical trials for stroke patients. Deviating from task-specific evaluations, the mRS measures the level of independence on a scale of 0 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Tadeja Hernja Rumpf, Principal Investigator — University Medical Centre Maribor, Slovenia
Locations (1):
- University Medical Centre Maribor, Ljubljanska 5 Maribor, Slovenia, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the small sample size and increased re-identification risk under GDPR. Aggregate results, study protocol, and statistical analysis plan will be made available upon publication.

REFERENCES:
- See also: Related Info — https://www.ukc-mb.si